CLINICAL TRIAL: NCT05183906
Title: Evaluation of Next-Generation Sequencing-based Metabarcoding Versus Culturing in Infectious Keratitis
Brief Title: Evaluation of Next-Generation Sequencing-based Metabarcoding Versus Culturing for Microbiological Assessment in Infectious Keratitis
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders Ivarsen, Consultant, Associate Professor, Aarhus University Hospital
Other Study IDs: KeratitisMicrobiome
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Keratitis
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — Evaluation of microbiological culturing versus next generation sequencing for ribosomal DNA

SUMMARY:
Infectious keratitis is a potential sight threatening condition. In conventional clinical practice culturing is performed in order to identify the causative microbial organism; however in recent years Next Generation Sequencing for the presence of ribosomal DNA from bacteria, fungi, or amoeba has become available. The present study aims to compare conventional culturing with Next Generation Sequencing for identifying microorganism causing keratitis.

DETAILED DESCRIPTION:
Patients admitted with microbial keratitis to the department of ophthalmology at Aarhus University Hospital is evaluated with both conventional culturing at agar plates, broth culture, and Next Generation Sequencing for ribosomal DNA.

Only patients with a corneal infiltrate of a minimum of 2 mm or of 1 mm within the central 6 mm of the cornea will be included in the study.

Sampling includes two samples from the contralateral healthy eye to control for the patient's normal microbiome, evaluated with culturing in broth and with NGS.

From the infiltrate, samples include culturing on Sabouraud agar, chocolate agar, and blood agar, culturing in broth medium, and samples for NGS.

A total of 100 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a corneal infiltrate of minimum 2 mm in diameter or of 1 mm diameter within the central 6 mm of the cornea

Exclusion Criteria:

- Patients below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with keratitis admitted to tertiary ophthalmological unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of clinically relevant microorganisms identified using culture or next generation sequencing | 1 year
Comparison of clinically relevant identified microorganisms on a genus level | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No